CLINICAL TRIAL: NCT00045331
Title: Are the Proteomic Profiles of Serum and Urine Predictivefor Clinical Outcome After Definitive Radiotherapy for Localized Prostate Cancer? A Preliminary Cohort Study
Brief Title: Study in Predicting Outcome of Patients Undergoing Radiation Therapy for Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: CDR0000256868; NCI-02-C-0226; NCT00039806 (obsolete NCT alias)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2004-10

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Genetic: proteomic profiling

SUMMARY:
RATIONALE: Proteins found in blood and urine samples may help predict outcome and allow doctors to plan more effective treatment.

PURPOSE: Diagnostic trial to study blood and urine proteins in predicting treatment outcome in patients who are undergoing radiation therapy for prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Correlate serum and urine protein profiles collected before or after radiotherapy with clinical outcome in patients with prostate cancer.
* Identify protein profiles that can distinguish between patients with no evidence of disease and those with biochemical and/or clinical failure.
* Determine whether those serum proteomic profiles consistent with failure can be identified at early time points in the course of treatment and follow-up of these patients.

OUTLINE: Patients are stratified according to clinical outcome (prior to radiotherapy vs no evidence of disease vs biochemical failure vs clinical failure vs clinical outcome not yet determined).

Urine and blood specimens are collected from patients either before or after definitive radiotherapy. Samples are analyzed by surface-enhanced laser desorption and ionization time-of-flight mass spectrometry to develop proteomic patterns.

Results of proteomic profiles do not influence patient care.

PROJECTED ACCRUAL: A total of 150 patients (30 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer
* Completed or planned definitive radiotherapy

PATIENT CHARACTERISTICS:

Age

* Adult

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Concurrent immunotherapy allowed

Chemotherapy

* Concurrent chemotherapy allowed

Endocrine therapy

* Concurrent hormonal therapy allowed

Radiotherapy

* See Disease Characteristics
* Concurrent palliative radiotherapy allowed

Surgery

* No prior prostatectomy, including radical prostatectomy
* No concurrent radical prostatectomy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-08; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Camphausen, MD, Study Chair — NCI - Radiation Oncology Branch; ROB
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland